CLINICAL TRIAL: NCT04048798
Title: Effect of Nasal High Flow on Perioperative Oxygenation in Patients Undergoing Bariatric Surgery
Brief Title: Nasal High Flow in Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr Cigdem Akyol Beyoğlu, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 88298
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; bariatric surgery; high frequency nasal cannula; oxygenation
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen therapy via HFNC (Active Comparator): Patients who will be applied high frequency nasal cannula before and after surgery
  Interventions: Other: Oxygen therapy via HFNC
- Oxygen therapy via face mask (Active Comparator): Patients who will be applied O2 via face mask before and after surgery
  Interventions: Other: Oxygen therapy via face mask

INTERVENTIONS:
Other: Oxygen therapy via HFNC — Oxygen treatment will be applied to the patients via HFNC before and after surgery
  Arms: Oxygen therapy via HFNC
Other: Oxygen therapy via face mask — Oxygen treatment will be applied to the patients via face mask before and after surgery
  Arms: Oxygen therapy via face mask

SUMMARY:
High frequency nasal cannula (HFNC) provides an inspiration O2 fraction of 21-1% and it has a minimal dead space and can be well tolerated due to humidified air. Group I patients will be applied HFNC before and after bariatric surgery, Group II patients will be applied a constant O2 concentration via face mask. Oxygen pressure, oxygen saturation, carbon dioxide, respiration frequency, forced vital capacity will be measured before and after surgery.

DETAILED DESCRIPTION:
Morbid obese patients are prone to atelectasis and hypoxemia after bariatric surgery. High frequency nasal cannula (HFNC) provides an inspiration O2 fraction of 21-1% and it has a minimal dead space and can be well tolerated due to humidified air. It provides 5-7 cm H2O positive end expiratory pressure to the airways and may prevent atelectasis. In the preoperative room, forced vital capacity, peripheral oxygen saturation (SpO2), respiratory frequency, heart rate (HR), blood pressure (BP), carbon dioxide, oxygen pressure and carbon dioxide partial pressure values in blood gas analysis will be recorded. We will apply HFNC in the preoperative and postoperative period to Group I patients, while applying a constant O2 concentration to Group II patients. After appliying HFNC for two hours in Group I patients and O2 via face mask in Group II patients measurements will be repeated. During surgery, similar mechanical ventilation parameters will be applied to the patients. After the operation Group I patients will be applied HFNC, while Group II patients will be applied O2 via face mask in the recovery room for two hours. Measurements will be repeated. Primary end point of the study is the association between oxygen pressure, carbon dioxide partial pressure values among preoperative before and after HFNC and O2 and postoperative times.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a body mass index of 40-55 kg/m2
* American Society of Anesthesiologists score II-III
* Patients undergoing laparoscopic sleeve gastrectomy or one anastomosis gastric bypass

Exclusion Criteria:

* Obstructive sleep apnea syndrome
* Using a non invasive mechanical ventilation device preoperatively
* Patients whoo will predicted to postanesthesia care unit admission postoperatively

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
PO2 value | 24 hours
  PO2 value will be measured before HFNC or face mask, after HFNC or face mask and after surgery
PCO2 value | 24 hours
  PO2 value will be measured before HFNC or face mask, after HFNC or face mask and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cigdem A BEYOGLU, Principal Investigator — İstanbul Üniversitesi- Cerrahpaşa Cerrahpaşa Tıp Fakültesi

IPD SHARING:
Plan to Share IPD: No
I am unaware of the advantages or disadvantages of sharing IPD

REFERENCES:
- [Background] Baraka AS, Taha SK, Siddik-Sayyid SM, Kanazi GE, El-Khatib MF, Dagher CM, Chehade JM, Abdallah FW, Hajj RE. Supplementation of pre-oxygenation in morbidly obese patients using nasopharyngeal oxygen insufflation. Anaesthesia. 2007 Aug;62(8):769-73. doi: 10.1111/j.1365-2044.2007.05104.x. PMID 17635423